CLINICAL TRIAL: NCT03959670
Title: Anatomical Feasibility of the Off-the-shelf E-nside Multibranch Stent Graft System (JOTEC GmbH, Hechingen) for Thoracoabdominal and Para-renal Aortic Aneurysms. (E-nside Study)
Brief Title: Anatomical Feasibility of the Off-the-shelf E-nside Multibranch Stent Graft System for Thoracoabdominal and Para-renal Aortic Aneurysms.(E-nside Study)
Acronym: E-nside
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Bertoglio Luca, Principal Investigator, IRCCS San Raffaele
Other Study IDs: E-nside study
Record Dates: First submitted 2019-05-16; First posted 2019-05-22 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Aortic Aneurysm, Thoracoabdominal; Para-renal Aortic Aneurysms
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- extensive TAAA: including Crawford extent I and II TAAA
- Crawford extent III TAAA
- supra-renal aortic aneurysms: Crawford extent IV TAAA and para-renal abdominal aortic aneurysms.

SUMMARY:
The study was created to evaluate the theoretical anatomical feasibility of the new E-nside Multibranch Stent Graft System (JOTEC GmbH, Hechingen) in patients with thoracoabdominal and para-renal aortic aneurysms based on retrospective review of pre-operative imaging studies of the patients treated with other techniques for this pathology in the vascular Unit of San Raffaele Hospital, in the past ten years. With this study, investigators want to analyze in how many cases the new prosthesis would be usable.

E-nside Multibranch Stent Graft System (JOTEC GmbH, Hechingen) is in the pre-CE marking stage. At present, the certifying organism is evaluating the documentation for the release the CE mark certification and Declaration of Conformity.

ELIGIBILITY:
Inclusion Criteria:

- patient who underwent treatment of thoracoabdominal or para-renal aortic aneurysm at San Raffaele Hospital between January 2007 and January 2017.

Exclusion Criteria:

- incomplete or inappropriate imaging quality defined as pre-operative CTAs with slice thickness >1-mm.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with thoracoabdominal or para-renal aortic aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 562 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Multi-planar and curved reconstruction of pre-operative contrast-enhanced computed tomography scans (CTA) | between January 2007 and January 2017
  Number of patients (already treated in the Vascular Surgery Unit of San Raffaele Hospital) with anatomical characteristic for use (theoretic)of the new E-nside Multibranch Stent Graft System.

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chuter TA, Rapp JH, Hiramoto JS, Schneider DB, Howell B, Reilly LM. Endovascular treatment of thoracoabdominal aortic aneurysms. J Vasc Surg. 2008 Jan;47(1):6-16. doi: 10.1016/j.jvs.2007.08.032. Epub 2007 Nov 5. PMID 17980540
- [Result] Sobocinski J, d'Utra G, O'Brien N, Midulla M, Maurel B, Guillou M, Azzaoui R, Roeder B, Resch TA, Haulon S. Off-the-shelf fenestrated endografts: a realistic option for more than 70% of patients with juxtarenal aneurysms. J Endovasc Ther. 2012 Apr;19(2):165-72. doi: 10.1583/11-3772.1. PMID 22545880
- [Derived] Bilman V, Cambiaghi T, Grandi A, Carta N, Melissano G, Chiesa R, Bertoglio L. Anatomical feasibility of a new off-the-shelf inner branch stent graft (E-nside) for endovascular treatment of thoraco-abdominal aneurysms. Eur J Cardiothorac Surg. 2020 Dec 1;58(6):1296-1303. doi: 10.1093/ejcts/ezaa276. PMID 33057585